CLINICAL TRIAL: NCT02376686
Title: Musik Als Nicht-pharmakologische Intervention Zur Behandlung Von Schlafstörungen Bei Patienten Mit Depressiven Erkrankungen
Brief Title: Music Intervention in the Treatment of Sleep Disorders for Depressed Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sanatorium Kilchberg AG (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KEK-ZH-Nr.2013-0544
Record Dates: First submitted 2014-08-26; First posted 2015-03-03 (Estimated); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Insomnia; Depression
Keywords: sleep Quality; Depression; Music; quality of life
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Music intervention (Experimental): Patient receives Music Intervention before going to sleep.
  Interventions: Other: Music intervention
- treatment as usual (No Intervention): Patient receives Treatment as usual.

INTERVENTIONS:
Other: Music intervention — Patient receives Music Intervention before going to sleep. It is composed Music which the Patient hear with maysound Music player.
  Arms: Music intervention

SUMMARY:
The purpose of this study is to determine whether music hearing in the evening before going to sleep can improve sleep quality, depressive symptoms and quality of life in patients with affective disorders.

DETAILED DESCRIPTION:
Disrupted sleep including Problems of initiating and maintaining sleep are most often symptoms in patients with depressive Syndromes and often persist after successful treatment of affective symptoms. Normally disrupted sleep in the context of affective disorder is treated with sleep medication, which can lead to severe and sometimes intolerable side effects.

A non-pharmacological approach for improving sleep Quality is Hearing Music before going to sleep. Classical indian Music can improve sleep Quality in depressed patients. In a danish study protocol Western Music improved sleep quality in patients with disturbed sleep and posttraumatic stress disorder.

The investigators want to use western Music to improve sleep . In a three week Intervention time, patients shall hear before going to sleep every night for one hour relaxing Music. The control group receives Treatment as usual. After the end of Intervention, every participant has the possibility to use the sleep inducing Music.

The aim of the study is to prove whether Hearing Music before going to sleep over three weeks improves subjective sleep quality, self rated depressive symptoms and Quality of life and objective Parameters such as sleep duration and sleep latency, measured by actigraphy. In a follow-up interview four weeks after the Intervention the investigators want to prove if the effects continue after end of Intervention.

ELIGIBILITY:
Inclusion Criteria:

* inpatient and outpatient treatment in Sanatorium Kilchberg
* one of the following diagnoses according to ICD 10: F32, F33, F34.1, F34.21, F34.8,
* Age between 18 and 65 years
* completed Primary education Level
* good command of the german language
* able to understand Patient information,
* given informed consent,

Exclusion Criteria:

* no informed consent
* one or more of the following diagnoses according to ICD 10: F32.3, F33.2, F31.3, F31.4, F60.31, F10, F13, F00, F01, F02, F03, G47.3, G25.8, H90, H91
* patients with acute suicidal tendency
* pregnant or breastfeeding women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-04; Primary Completion 2023-02 (Actual); Study Completion 2023-02 (Actual)

PRIMARY OUTCOMES:
objective sleep Quality | up to four weeks
  Measurement with actimeter

SECONDARY OUTCOMES:
subjective sleep Quality | up to eight weeks
  Measurement by questionnaire, Pittsburg Sleep Quality Index

OTHER OUTCOMES:
severity of depressive symptoms | up to eight weeks
  Measurement by questionnaire, Beck Depression inventory

CONTACTS AND LOCATIONS:
Overall Officials: Katja Cattapan, MD, Principal Investigator — Sanatorium Kilchberg AG
Locations (1):
- Sanatorium Kilchberg AG, Kilchberg, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
Partial availability is possible

REFERENCES:
- [Background] Jespersen KV, Vuust P. The Effect of Relaxation Music Listening on Sleep Quality in Traumatized Refugees: A Pilot Study. J Music Ther. 2012 Summer;49(2):205-29. doi: 10.1093/jmt/49.2.205. PMID 26753218
- [Background] Maratos AS, Gold C, Wang X, Crawford MJ. Music therapy for depression. Cochrane Database Syst Rev. 2008 Jan 23;(1):CD004517. doi: 10.1002/14651858.CD004517.pub2. PMID 18254052
- [Background] Jindal RD, Thase ME. Treatment of insomnia associated with clinical depression. Sleep Med Rev. 2004 Feb;8(1):19-30. doi: 10.1016/S1087-0792(03)00025-X. PMID 15062208
- [Background] Harmat L, Takacs J, Bodizs R. Music improves sleep quality in students. J Adv Nurs. 2008 May;62(3):327-35. doi: 10.1111/j.1365-2648.2008.04602.x. PMID 18426457
- [Derived] Jespersen KV, Pando-Naude V, Koenig J, Jennum P, Vuust P. Listening to music for insomnia in adults. Cochrane Database Syst Rev. 2022 Aug 24;8(8):CD010459. doi: 10.1002/14651858.CD010459.pub3. PMID 36000763